CLINICAL TRIAL: NCT07244146
Title: Effects of Comprehensive Hand Intense Strength Training on In Hand Manipulation and Grip Strength Among Children With Spastic Cerebral Palsy
Brief Title: Effects of CHRIST Among Children With Spastic CP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: REC/RCR&AHS/FAIRY ALI
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Cerebral Palsy
Keywords: Hemiplegic spastic cerebral palsy; In-hand manipulation; , Grip strength
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: This Quasi experimental study investigates the effects of CHRIST on In Hand Manipulation and Grip Strength amonfg children with Spastic Cerebral Palsy. The study involves 14 children from 6-12 years of age, and will be given intervention for 10 weeks period.
  Key performance outcomes- In Hand Manipulation and Grip Strength will be assessed both before and after the intervention. This study aims to address this gap by evaluating the effects of the CHRIST on IHM and grip strength in children diagnosed with spastic cerebral palsy. The hypothesis is that integrating strength training with high repetition, functionally relevant tasks yields greater and more practical gains than strength training or conventional therapy alone. Data will be analyzed through SPSS version 27.0
Masking Description: Single (Participant) Participants will get separate treatment protocols and possible efforts will be put to mask the both group about the treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The intervention will be comprehensive hand repetitive intense strength training (Experimental): CHRIST, is a treadmill-based training with body weight supported by the upper limbs. There will be a session of 40 minutes, which includes 3 sets (10 minutes exercise with 3 minutes rest period per set), three times a week, over a 10 week period. By maintaining the posture of the quadruped, the abdomen and weight of the lower limb will be supported by using a support board under the abdomen. The speed of the treadmill for the upper limbs will be 0.3-1.2 km/h. Results will be evaluated by MA2 and dynamometer.
  Interventions: Other: CHRIST

INTERVENTIONS:
Other: CHRIST — CHRIST, is a treadmill-based training with body weight supported by the upper limbs. There will be a session of 40 minutes, which includes 3 sets (10 minutes exercise with 3 minutes rest period per set), three times a week, over a 10 week period. By maintaining the posture of the quadruped, the abdomen and weight of the lower limb will be supported by using a support board under the abdomen. The speed of the treadmill for the upper limbs will be 0.3-1.2 km/h.

SUMMARY:
This Quasi experimental study investigates the effects of CHRIST on In Hand Manipulation and Grip Strength amonfg children with Spastic Cerebral Palsy. The study involves 14 children from 6-12 years of age, and will be given intervention for 10 weeks period.

Key performance outcomes- In Hand Manipulation and Grip Strength will be assessed both before and after the intervention. This study aims to address this gap by evaluating the effects of the CHRIST on IHM and grip strength in children diagnosed with spastic cerebral palsy. The hypothesis is that integrating strength training with high repetition, functionally relevant tasks yields greater and more practical gains than strength training or conventional therapy alone. Data will be analyzed through SPSS version 27.0

DETAILED DESCRIPTION:
This Quasi Experimental study investigates the effects of CHRIST on In Hand Manipulation and Grip Strength in children with Spastic Cerebral Palsy. CHRIST was designed to enhance the motor ability of children. The efficacy of this program will be investigated through a Quasi Experimental study. Data will be collected from special schools and rehabilitation centers having children with spastic cerebral palsy. The intervention CHRIST will be given thrice a week for forty minutes. The study will be completed in 10 weeks after approval of the synopsis. The study will include 14 children, male and female. Inclusion criteria for the study will include patients diagnosed with spastic CP. Data will be collected from children aged 6 to 12 years old. IHM will be measured by Melbourne Assessment 2 scale (MA2). Grip Strength will be measured by dynamometer. IHM & Grip Strength will be assessed both before and after the intervention.This study aims to address this gap by evaluating the effects of CHRIST on IHM and grip strength in children diagnosed with spastic cerebral palsy. The hypothesis is that integrating strength training with high repetition, functionally relevant tasks yields greater and more practical gains than strength training or conventional therapy alone. Data will be analyzed through SPSS version 27.0

ELIGIBILITY:
Inclusion Criteria:

* Children Diagnosed with hemiplegic spastic cerebral palsy.
* Age 6-12 years.
* Capable of following commands regarding hand use and testing.
* Capable of communicating needs.
* Parents or caregivers willing to provide informed consent and participate in the study.
* No contraindications to moderate physical activity.
* Able to lift the more affected arm 15 cm above a table surface and grasp light objects

Exclusion Criteria:

* Children with musculoskeletal system injuries, including upper limb fractures or contractures, as well as those who had received medications affecting muscle strength or spasticity, were excluded from the study.
* Orthopedic surgery involving the more affected hand within the past 6 months.
* Children with Cardiovascular disease.
* Lack of cooperation with instructions or other behavioral challenges that prevent effective delivery of intensive therapy.
* Visual impairments that may hinder active participation.
* Seizure or family history of seizure disorders

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Estimated)
Dates: Start 2025-10-22 (Actual); Primary Completion 2026-06-02 (Estimated); Study Completion 2026-06-16 (Estimated)

PRIMARY OUTCOMES:
Jamma Dynamometer | Baseline, 1st week and 10th week
  Grip strength will be measured by Jammar Dynamometer. The hand-held dynamometer are reliable measurement instruments to measure muscle strength of the arm and hand in children with unilateral spastic cerebral palsy, aged 7 12 years

SECONDARY OUTCOMES:
Melbourne assessment 2 (MA2) | Baseline, 1st week and 10th week
  Melbourne Assessment 2 (MA2) will be used to assess in-hand manipulation before and after the intervention (CHRIST) to evaluate the impact. MA2 is a reliable and valid tool for assessment of upper limb in children with CP.

CONTACTS AND LOCATIONS:
Overall Officials: FAIRY ALI, MSPT, Principal Investigator — Riphah International University
Locations (1):
- Imran Amjad, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee DR, You JH, Lee NG, Oh JH, Cha YJ. Comprehensive Hand Repetitive Intensive Strengthening Training (CHRIST)-induced morphological changes in muscle size and associated motor improvement in a child with cerebral palsy: an experimenter-blind study. NeuroRehabilitation. 2009;24(2):109-17. doi: 10.3233/NRE-2009-0460. PMID 19339750